CLINICAL TRIAL: NCT05080530
Title: Vitamin D (200 000 IU) for the Treatment of Painful Diabetic Neuropathy
Brief Title: Vitamin D and Painful Diabetic Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baqai Institute of Diabetology and Endocrinology (Other)
Collaborators: Scotmann Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Abdul Basit, Professor of Medicine, and Director, Baqai Institute of Diabetology and Endocrinology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIDE-216D/2021
Record Dates: First submitted 2021-09-29; First posted 2021-10-15 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Painful Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1. Normal Vit D (> 30ng/mL) (No Intervention): Follow-up after 3 months with standard treatment
- 2. Insufficient Vit D (20-30ng/mL) (Experimental): single oral dose capsule 200,000 IU of Cholecalciferol
  Interventions: Drug: Cholecalciferol
- 3. Insufficient Vit D (20-30ng/mL) (No Intervention): Follow-up after 3 months with standard treatment
- 4. Deficient Vit D (Experimental): single oral dose capsule 200,000 IU of Cholecalciferol
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — Effect of Vitamin D on diabetic neuropathy symptoms
  Other Names: Sunny D™ (Vitamin D3) Softgel Capsule
  Arms: 2. Insufficient Vit D (20-30ng/mL); 4. Deficient Vit D

SUMMARY:
The main objective of this study is to evaluate the effect of vitamin D3 on diabetic individual with painful neuropathy in a tertiary healthcare.

The people with diabetes (type 1 and type 2) who have a Douleur Neuropathique 4 (DN4) score ≥4 will be considered eligible in this prospective study. Their serum samples will be subjected to pre-and post-biochemical screening of serum 25 (OH) D and HbA1c. The individual having Vitamin D insufficiency and deficiency will be administered a single dose of oral Vitamin D3 (Soft Gel capsule 200,000 IU), and follow-up for post-biochemical screening after 3 months.

DETAILED DESCRIPTION:
Painful diabetic neuropathy (PDN) is the most common diabetic complication in patients who have had diabetes mellitus for a long time. Diabetic peripheral neuropathy is the common cause of neuropathy globally. About 50-60% of individuals with long-term diabetes develop diabetic neuropathy. Several recent observational studies in diabetic individuals have provided a correlation between vitamin D insufficiency and diabetes. Despite the fact that the pathogenesis of diabetic neuropathy is complex, recent investigations revealed that deficiency of vitamin D is an important factor in the development of diabetic neuropathy. Also, vitamin D supplementation was found to be effective in treating neuropathic pain and preventing neuronal degeneration.

Aims and Objectives:

The assessment of the effect of single-dose, oral vitamin D in patients with painful diabetic neuropathy.

Materials and Methods:

Study Drug: Oral cholecalciferol (Vitamin D3 capsule 200,000 IU).

A single oral dose of 200000 IU vitamin D will be administered in people with diabetic neuropathy, and the effect will be observed after 3 months.

* Sample size = 216 type 1 and 2 diabetic subjects
* Recruitment time = 4 months
* Treatment duration = 3 months

Ethical Approval:

The ethical approval for this study will be taken from the Institutional Review Board (IRB) of Baqai Institute of Diabetology and Endocrinology (BIDE)

Study Area and Duration:

This study is going to be conducted from October 2021 to March 2022 in the outpatient department (OPD) of BIDE.

Data Analysis and Statistics:

The primary analysis will compare the change from baseline. Comparisons within each treatment group across time will also be considered. The analysis will be performed with the Statistical Package for the Social Sciences (SPSS).

Assessment during the Treatment Period:

* Change from baseline in DN4
* Change from baseline in serum 25 (OH) D,
* Change from baseline in HbA1c

ELIGIBILITY:
Inclusion Criteria:

* Insulin dependent diabetes
* Insulin independent diabetes
* Age range between 25 to 80 years
* Glycated hemoglobin (HbA1c) level must be ≥ 6.5%
* Apparently no symptoms of Vitamin D Deficiency

Exclusion Criteria:

* History of hyperparathyroidism
* Pregnant women
* Lactating mothers
* History for rickets and osteomalacia
* On Vitamin D supplementation
* On Multivitamin
* On anti-epileptics
* On steroids
* On bisphosphonates
* On oral contraceptives
* Subjects who refuse to participate in the study

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2021-10-29 (Actual); Primary Completion 2022-08-20 (Estimated); Study Completion 2022-08-20 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in DN4 score. | 3 months
  The change will be observed with the help of neuropathic pain assessment questionnaire.
Change from baseline in serum HbA1c. | 3 months
  The change will be observed in the serum values of glycated hemoglobin at the end point after the administration of vitamin D.
Change from baseline in serum vitamin D. | 3 months
  The cholecalciferol (Vitamin D) level in serum will be observed at the end point after the administration of vitamin D.

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Basit, Director, Principal Investigator — Baqai Institute of Diabetology and Endocrinology (BIDE)
Locations (1):
- Baqai Institute of Diabetology and Endocrinology (BIDE), Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No